CLINICAL TRIAL: NCT06779435
Title: A Multicenter, Prospective, Real-world Study of a Regimen Containing Tucidinostat for Primary Treatment of Diffuse Large B-cell Lymphoma
Brief Title: A Multicenter, Prospective, Real-world Study of a Regimen Containing Tucidinostat for Primary Treatment of DLBCL
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Principal Investigator, Ruijin Hospital
Other Study IDs: CSIIT-B42
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: DLBCL
Keywords: Tucidinostat; DLBCL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: DLBCL patients diagnosed unfit/ Unfit.: A person who is unfit/ unfit is defined as being 80 years or older, or younger than 80 years old but has comorbidities and cannot tolerate a standard dose of chemotherapy as determined by the investigator.
  Interventions: Drug: Low intensity treatment options
- Cohort 2: Patients diagnosed with DLBCL who cannot be classified as unfit/ Unfit.: Cohort 2: Patients diagnosed with DLBCL who cannot be classified as unfit/ Unfit.
  Interventions: Drug: Conventional immunochemotherapy regimen

INTERVENTIONS:
Drug: Low intensity treatment options — Reference options for a combined regimen include C-R2, C-R-mini-CHOP, etc.
  Subjects whose efficacy is assessed as CR after the end of induction therapy will enter consolidation therapy. Tucidinostat maintenance therapy or autologous hematopoietic stem cell transplantation may be an option. Tucidinostat maintenance therapy will be performed every 3 weeks. .Single-drug maintenance is recommended to last 24 weeks
  Groups: Cohort 1: DLBCL patients diagnosed unfit/ Unfit.
Drug: Conventional immunochemotherapy regimen — Reference options for a combined regimen include CR-CHOP, C-Pola-R-CHP, etc.
  Subjects whose efficacy is assessed as CR after the end of induction therapy will enter consolidation therapy. Tucidinostat maintenance therapy or autologous hematopoietic stem cell transplantation may be an option. Tucidinostat maintenance therapy will be performed every 3 weeks. Single-drug maintenance is recommended to last 24 weeks
  Groups: Cohort 2: Patients diagnosed with DLBCL who cannot be classified as unfit/ Unfit.

SUMMARY:
This is a prospective, observational, multicenter, cohort study with 400 newly treated DLBCL patients. To evaluate the clinical efficacy and safety of tucidinostat in the real-world treatment of primary diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
The study was divided into 2 cohorts. Cohort 1: DLBCL patients diagnosed unfit/ Unfit. A person who is unfit/ unfit is defined as being 80 years or older, or younger than 80 years old but has comorbidities and cannot tolerate a standard dose of chemotherapy as determined by the investigator. Reference options for a combination regimen include C-R2, C-R-mini-CHOP, etc.

Cohort 2: Patients diagnosed with DLBCL who cannot be classified as unfit/ Unfit. Reference options for a combination regimen include CR-CHOP, C-Pola-R-CHP, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, male or female;
* 2. No previous treatment for DLBCL, including chemotherapy, targeted therapy and immunotherapy;
* 3. DEL [Diffuse large B-cell lymphoma with double expression of MYC and BCL2 (immunohistochemical MYC≥40%, BCL2≥50%)] was confirmed by pathology; Or non-double expression but at least one of the following:;

  1. TP53 or other epigenetic gene mutations (as in: ACTB, BCL6, BCOR, CREBBP, EP300, EZH2, HIST1H1C, HIST1H1E, HIST1H2BK, HIST2H2AB, IRF4, KMT2A, KMT2C, KMT2D, MYC, MYD88, NSD2, RAG1, SETD1B SF3B1, SIN3A, TBL1XR1, TET2, TOX, TP53, TRIP12, TRRAP, UBE2A)
  2. MYC and BCL2 double hit
* 4. Plan to receive or are receiving a treatment regimen containing tucidinostat (if it is permitted to start using tucidinostat after obtaining specific test results due to pending genetic sequencing results);
* 5. Voluntarily sign informed consent.

Exclusion Criteria:

* 1. Patients currently enrolled or planning to participate in any interventional clinical trial;
* 2. The expected survival time is less than 6 months;
* 3. There are any other reasons that the investigators believe are not suitable for patients to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
EFS（Event-free survival） | 2-year
  The length of time from the start of treatment to the onset of disease progression, recurrence after CR, death from any cause, or the start of new therapy for residual lesions (including conversion therapy for lesions during the trial) after the end of combination therapy, whichever occurs first.

SECONDARY OUTCOMES:
CRR（Complete response rate） | End of treatment visit (6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  The number of subjects who achieved complete response (CR) at the end of combination therapy as a percentage of the total number of participants in the analysis.
PFS（Progression-free survival） | 2-year
  The length of time from the start of treatment to the onset of disease progression or recurrence or death from any cause, whichever occurs first
OS（Overall survival） | 2-year
  From the start of treatment to the time of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 197 Ruijin 2nd Road, Huangpu District, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No